CLINICAL TRIAL: NCT01091649
Title: An Open-label, Randomized, Crossover Study to Evaluate the Bioavailability of Two Candidate Tablet Formulations of ABT-450 With Reference to the Hard Gelatin Capsule Formulation
Brief Title: Study in Healthy Adults to Evaluate the Bioavailability of Two Test Tablet Formulations of ABT-450
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Adebayo Lawal, Global Project Director, Abbott
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: M10-797
Record Dates: First submitted 2010-02-26; First posted 2010-03-24 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Pharmacokinetics, Safety
MeSH Terms: interventions — paritaprevir; Ritonavir

ARMS (5):
- A (Active Comparator): Low dose ABT-450 capsule and ritonavir capsules (reference).
  Interventions: Drug: ABT-450; Drug: ritonavir
- B (Active Comparator): Low dose ABT-450 SDD Tablet Form 1 and ritonavir capsules (test 1)
  Interventions: Drug: ABT-450; Drug: ritonavir
- C (Active Comparator): Low dose ABT-450 SDD Tablet Form 2 and ritonavir capsules (test 2).
  Interventions: Drug: ABT-450; Drug: ritonavir
- D (Active Comparator): High dose ABT-450 capsule and ritonavir capsules (reference).
  Interventions: Drug: ritonavir; Drug: ABT-450
- E (Active Comparator): High dose ABT-450 SDD Tablet Form 1 or 2 and ritonavir capsule (test)
  Interventions: Drug: ritonavir; Drug: ABT-450

INTERVENTIONS:
Drug: ABT-450 — Low dose ABT-450 / ritonavir see Arm Description for more information
  Arms: A; B; C
Drug: ritonavir — ritonavir see Arm Description for more information
  Other Names: ABT-538, ritonavir, Norvir
Drug: ABT-450 — High dose ABT-450 / ritonavir See Arm Description for more information
  Arms: D; E

SUMMARY:
The objective of this study is to assess the relative bioavailability of two test tablet formulations of ABT-450 as compared to the ABT-450 hard gelatin capsule formulation as a reference.

DETAILED DESCRIPTION:
This is a two part study. Part 1 is a single dose, three period, complete crossover study in approximately 21 subjects. Part 2 is a single dose, two period, complete crossover study in approximately 20 subjects.

ELIGIBILITY:
Inclusion Criteria

* Overall healthy subjects
* Non-childbearing potential females included

Exclusion Criteria

* Positive test for HAV IgM, HBsAg, anti-HCV Ab or anti-HIV Ab
* Clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder
* Use of tobacco or nicotine-containing products with the 6-month period prior to study drug administration
* Abnormal screening laboratory results that are considered clinically significant by the investigator
* Pregnant or breastfeeding female; requirement for any OTC and/or prescription medication, vitamins and/or herbal supplements on a regular basis
* Previous exposure to ABT-450

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Assessment of Pharmacokinetics of two ABT-450 tablet formulations plus ritonavir and the ABT-450 capsule formulation plus ritonavir. Each dosed at low ABT-450/ritonavir | 72 hrs post dose
Assessment of Pharmacokinetics of the selected ABT-450 tablet formulations plus ritonavir and the ABT-450 capsule formulation plus ritonavir. Each dosed at high ABT-450/ritonavir | 72 hrs post dose

SECONDARY OUTCOMES:
To tabulate treatment emergent adverse events of two ABT-450 tablet formulations plus ritonavir and the ABT-450 capsule formulation plus ritonavir | Through 30 days post last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Adebayo Lawal, M.D., Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 27781, Waukegan, Illinois, United States